CLINICAL TRIAL: NCT04657432
Title: Accelerated Repetitive TMS for Affective Dysfunction: Establishing the Dose-Response Curve
Brief Title: Brief, High-dose rTMS for Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00084111
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Study 1: Participants will be randomized to 10 different doses of accelerated intermittent theta burst rTMS for remediation of depression symptoms. The goal is to determine the optimal dose in terms of efficacy while minimizing burden and side effects.
  Study 2: Participants will be assigned to 10 active sessions (per treatment day) of accelerated rTMS for 5 treatment days. All doses are active and within established therapeutic levels of rTMS. The goal is to determine the role of individual variations of their functional networks compared to the site of stimulation.
Who Masked: Participant
Masking Description: Study 1: All participants will be randomized to 10 different active doses of accelerated, intermittent theta burst rTMS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (11):
- Dose 1 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is five sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 2 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 2 is 10 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 3 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 3 is 15 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 4 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 4 is 20 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 5 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 5 is 20 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 6 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 6 is 25 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 7 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 7 is 30 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 8 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 8 is 35 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 9 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 9 is 40 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Dose 10 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 10 is 40 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Study 2: 10 Active Doses (Experimental): All participants will be assigned to 10 sessions (per treatment day) of accelerated rTMS for 5 treatment days. All doses are active and within established therapeutic levels of rTMS. Dose 10 is 50 active sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — MagVenture MagPro TMS System would be utilized to deliver 3-minute sessions of intermittent theta burst to left dorsolateral prefrontal cortex.

SUMMARY:
High frequency repetitive transcranial magnetic stimulation (rTMS) has been shown to be safe, feasible, and acceptable. Conventionally, rTMS investigations have relied on rational decision trees for dosage determination. The purpose of this study is to systematically examine an accelerated protocol of intermittent theta burst (iTBS). Study 1 aims to provide a quantifiable dose-response curve for iTBS and depressive symptom reduction in major depression. Study 2 aims to determine the role of individual variations of their functional networks compared to the site of stimulation and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A negative urine pregnancy test, if female subject of childbearing potential.
* Able to speak English and complete study forms, adhere to treatment regimens, and be willing to return for regular visits.
* After full explanation of the study, willingness of participant is demonstrated by signing the informed consent form.

Exclusion Criteria:

* Clinically unstable medical disease:

  * cardiovascular
  * renal
  * gastrointestinal
  * pulmonary
  * metabolic
  * endocrine
  * other
* CNS disease deemed progressive
* Moderate or severe traumatic brain injury (TBI)
* Pregnant females or those currently breast-feeding.
* Current or history of schizophrenia or other psychotic disorder, except psychosis not otherwise specified (NOS) when the presence of sensory hallucinations is clearly related to the subject's trauma, Bipolar Type I disorder, or dementia:

  * vascular
  * Alzheimer's disease
  * other types
* Repeated abuse or dependence upon drugs (excluding nicotine and caffeine) within 6 days of study entry, with the exception of alcohol use disorder, which, at the discretion of the study team, may be permitted.

See further explanation under protection from risk.

* Active participation or plan for enrollment in another evidence-based psychotherapeutic clinical trial
* Participation in other psychotherapeutic modalities must have been stable for 3 months prior to enrollment and must remain stable throughout participation.
* Currently taking medications that have short half-lives, lower the seizure threshold, and do not have evidence of antidepressant efficacy. These include:

  * high dose theophylline or stimulants such as methylphenidate patients taking bupropion must be on a stable dose and take less than or equal to 300 mg/day. Stable means the same dose for 5 half-lives.
* An implanted device in subject's head (shunt, cochlear implant) and/or metal in subject's head (other than dental implant).
* History of seizures or a seizure disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Depression severity (change in score) | Day 1, post-treatment point of 1 month
  Depression severity as assessed by:
  1. Hamilton Scale for Depression (HAM-D) Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. 10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe.
Depression severity (change in score) | Day 1, post-treatment point of 1 month
  Depression severity as assessed by:
  2. Montgomery-Asberg Depression Rating Scale (MADRS) Rating lies on the defined scale steps (0, 2, 4, 6) or between them (1, 3, 5). Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.
Depression severity (change in score) | Day 1, post-treatment point of 1 month
  Depression severity as assessed by:
  3. Beck Depression Inventory-II (BDI-II) Rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63.

SECONDARY OUTCOMES:
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  1. Inventory of Depression and Anxious Symptoms (IDAS-II)
  -Questions are rated on a scale from 1-5 and covers a wide array of psychological measures
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  2. Mood and Anxiety Symptom Questionnaire
  -Questions designed to assess symptoms of general distress using a 5-point Likert scale ranging from 1"not at all" to 5 "extremely".
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  3. Penn State Worry Questionnaire
  -Questions are rated on a scale from: 1-Not at all typical of me to 5-Very typical of me. Possible range of scores is 16-80 with the algorithm of Total scores: 16-39 Low Worry, 40-59 Moderate Worry, and 60-80 High Worry
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  4. PTSD Checklist (PCL-5)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including:
  Monitoring symptom change during and after treatment Screening individuals for PTSD Making a provisional PTSD diagnosis
  -Questions are rated on a 5-point Likert scale (0 = "Not at all" to 4 = "Extremely")
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  5. Life Events Checklist (LEC-5) The Life Events Checklist for DSM-5 (LEC-5) is a self-report measure designed to screen for potentially traumatic events in a respondent's lifetime. The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items.
  -Responses are as followed: Happened to me; Witnessed it; Learned about it; Part of my job; Not sure; Doesn't apply
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  6. Childhood Trauma Questionnaire
  -The Childhood Trauma Questionnaire is a brief survey of six early traumatic experiences (death, divorce, violence, sexual abuse, illness or other), and assesses individual's understanding of their childhood trauma.
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  7. Fagerstrom Test for Nicotine Dependence
  -Yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  8. Alcohol Use Disorders Identification Test (AUDIT)
  -The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviors, and alcohol-related problems.
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  9. World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
  -Questions are rated on a a 5 point scale (from 0-4) Likert scale
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  10. World Health Organization Quality of Life - Brief Form (WHOQOL-BF)
  -Questions are rated on a a 5 point scale (from 1-5) Likert scale
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  11. Illness Intrusive Rating Scale (IIRS)
  -Questions are rated on a a 7 point scale (from 1-7) Likert scale which is a measure of the psychosocial impact of chronic disease
Comorbid symptom severity, functional impairment, acceptability, and tolerability | Day 1, post-treatment point of 1 month
  Participants would complete various questionnaires (change in score assessed):
  12. Quality of Life and Enjoyment and Satisfaction Questionnaire -Short Form (Q-LES-Q-SF)
  -Questions are rated on a 5 point scale (from 1-5) Likert scale. The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04657432/ICF_002.pdf